CLINICAL TRIAL: NCT07195500
Title: the Clinical Application of Somatostatin Receptor and Norepinephrine Transporter Targeted Imaging for the Diagnosis and Staging of Neuroblastoma and Pheochromocytoma/Paraganglioma
Brief Title: Clinical Application of Somatostatin Receptor and Norepinephrine Transporter Targeted Imaging for Diagnosis and Staging of Neuroblastoma and Pheochromocytoma/Paraganglioma
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20250819-16
Record Dates: First submitted 2025-08-29; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Neuroblastoma; Pheochromocytoma; Paraganglioma
Keywords: neuroblastoma; PET; pheochromocytoma; paraganglioma; somatostatin receptor; norepinephrine transporter
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Peripheral blood: serum and plasma aliquots collected at imaging time points and/or routine safety labs; selected leftover whole blood in EDTA tubes may be retained for assay validation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuroblastoma and PPGL Patients Undergoing SSTR/NET Imaging: This cohort includes patients with suspected or confirmed neuroblastoma (NB) or pheochromocytoma/paraganglioma (PPGL) undergoing somatostatin receptor (SSTR) and/or norepinephrine transporter (NET)-targeted molecular imaging for diagnostic evaluation and staging. Interventions of interest are diagnostic radiopharmaceutical administrations followed by imaging-there is no therapeutic intent. Participants may receive one or more NET tracers, including 18F-MFBG, 123I-MIBG, 131I-MIBG (legacy diagnostic where appropriate), 18F-LMI1195, and/or SSTR tracers, including 68Ga-DOTATATE, 68Ga-DOTATOC, 68Ga-DOTANOC, 64Cu-DOTATATE, 18F-SiTATE, 18F-AlF-NOTA-octreotide, depending on clinical indication and site availability. Imaging is performed on PET/CT or PET/MRI for PET tracers and SPECT/CT for SPECT tracers using harmonized acquisition and reconstruction parameters. When clinically justified

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic efficacy of somatostatin receptor and norepinephrine transporter targeted imaging (including 18F-MFBG, 123I-MIBG, 131I-MIBG, 68Ga-DOTA-NOC, 68Ga-DOTA-TATE, 68Ga-DOTA-TOC, and other radiolabeled somatostatin analogues) in the diagnosis and staging of neuroblastoma and pheochromocytoma/paraganglioma patients aged 1-70 years. The main questions it aims to answer are:

Can molecular targeted imaging using various norepinephrine transporter tracers (18F-MFBG, 123I/131I-MIBG) and somatostatin receptor tracers (68Ga-DOTA-peptides series) accurately detect primary tumors and metastatic lesions in neuroblastoma/pheochromocytoma patients? What is the comparative diagnostic performance (sensitivity, specificity, accuracy) of different molecular imaging techniques compared to histopathological diagnosis as the gold standard? Researchers will compare the imaging findings from multiple tracer types with surgical pathology results to assess diagnostic accuracy and clinical staging precision.

Participants will:

* Undergo screening assessments including medical history, physical examination, and laboratory tests
* Receive intravenous injection of selected tracers (18F-MFBG, 68Ga-DOTA-NOC/TATE, or other appropriate agents) at standardized doses followed by PET-CT/MRI imaging at optimal time points
* Undergo histopathological examination within 2 months post-imaging
* Complete safety follow-up for 6 months to monitor for any adverse reactions to the imaging agents

DETAILED DESCRIPTION:
This single-center, open-label diagnostic imaging study investigates the clinical utility of somatostatin receptor (SSTR) and norepinephrine transporter (NET) targeted molecular imaging for detection, staging, and treatment planning in patients with neuroblastoma and pheochromocytoma/paraganglioma (PPGL). The biological rationale rests on the frequent overexpression of NET in sympathoneuronal tumors and SSTR in neuroendocrine-derived neoplasms, enabling high-contrast visualization of primary and metastatic disease, including bone and bone marrow involvement. The protocol emphasizes harmonized acquisition and reconstruction parameters, quantitative analysis, and rigorous comparison against a composite reference standard comprising histopathology when available and multidisciplinary clinical adjudication.

The imaging strategy purposefully includes a broad spectrum of tracers within the SSTR and NET classes to capture complementary biology and to accommodate variability in patient phenotype, prior therapies, and local availability. For NET-targeted imaging, the study may employ 123I-metaiodobenzylguanidine (123I-MIBG) with planar and SPECT/CT techniques, 131I-MIBG as a legacy diagnostic alternative where appropriate, 18F-meta-fluorobenzylguanidine (18F-MFBG) for PET/CT or PET/MRI with improved resolution and logistics, 18F-LMI1195 as an investigational PET agent subject to site availability, 11C-hydroxyephedrine (11C-HED) PET where a cyclotron is accessible, and 18F-fluorodopamine (18F-FDA) PET in centers with established protocols. For SSTR-targeted imaging, the protocol allows 68Ga-DOTATATE, 68Ga-DOTATOC, and 68Ga-DOTANOC PET/CT or PET/MRI as contemporary standards; 64Cu-DOTATATE to leverage its longer half-life and extended imaging window; 18F-labeled SSTR agents such as 18F-SiTATE and 18F-AlF-NOTA-octreotide where available; and legacy SPECT agents including 111In-pentetreotide (Octreoscan) and 99mTc-HYNIC-TOC or 99mTc-EDDA/HYNIC-TOC depending on local practice. Tracer selection is individualized based on clinical indication, age, renal and hepatic function, concomitant medications, and logistical factors; when clinically justified and feasible, intra-patient multi-tracer imaging within and across SSTR and NET classes may be performed to enable head-to-head comparisons.

FDG and CXCR4 PET/CT or PET/MRI may be performed solely as optional comparator imaging at investigator discretion and contingent on site capability and local approvals. Optional comparators include 18F-FDG and CXCR4-targeted agents such as 68Ga-Pentixafor (and 64Cu-Pentixafor where permitted). These scans are not required for enrollment or primary analyses but may support exploratory comparisons in predefined subgroups.

Radiopharmaceutical preparation follows good manufacturing practice with predefined batch release specifications, including radiochemical purity (typically ≥95% for PET peptides), acceptable pH range, sterility, endotoxin limits, and specific activity as applicable. Each batch is accompanied by a certificate of analysis, lot traceability, and temperature and transport documentation, and any deviations are handled under corrective and preventive action procedures. Handling, storage, and administration comply with institutional radiation safety policies and national regulations. For optional comparator agents, applicable pharmacopeial or investigator's brochure specifications are followed.

Patient preparation adheres to tracer-specific guidance. For NET imaging, medications that interfere with catecholamine transport or storage (for example, labetalol and certain antidepressants) are reviewed and managed per site standard operating procedures, and thyroid blockade is implemented when indicated for radioiodine-labeled agents. For SSTR imaging, somatostatin analogues are managed to minimize receptor blockade when clinically appropriate. Hydration and frequent voiding are encouraged to reduce background activity. When optional 18F-FDG imaging is performed, patients fast for at least 4-6 hours, non-glucose-containing hydration is encouraged, strenuous exercise is avoided for 24 hours, and blood glucose is checked and documented prior to injection; insulin correction, if used, follows site policy to avoid altered biodistribution. When optional CXCR4 imaging is performed, no specific dietary restrictions apply; recent exposure to hematopoietic growth factors (for example, G-CSF) is recorded, and imaging may be deferred when clinically safe to mitigate confounding marrow uptake.

Acquisition timing follows established windows, such as approximately 90-180 minutes post-injection for 18F-MFBG, about 20-24 hours for 123I-MIBG planar/SPECT-CT (with optional early or delayed views), roughly 45-90 minutes for 68Ga-DOTA-peptides, approximately 60-180 minutes for 64Cu-DOTATATE, and around 60-120 minutes for 18F-labeled SSTR agents. For optional comparator scans, the recommended uptake times are approximately 50-70 minutes for 18F-FDG (acceptable range 45-90 minutes, time-stamped) and approximately 45-75 minutes for 68Ga-Pentixafor. Whole-body coverage typically spans from the skull vertex to mid-thigh, extended as clinically indicated; PET imaging uses 3D acquisition with attenuation and scatter correction, and SPECT employs iterative reconstruction with CT-based attenuation and scatter correction when available. Pediatric protocols prioritize dose optimization and motion mitigation, including sedation per institutional policy when required.

Quantitative analysis uses standardized regions of interest to derive SUVmax and SUVmean for PET, lesion-to-background ratios, and optional volumetric metrics such as total lesion uptake and metabolic or receptor-expressing tumor volume. For SPECT, semi-quantitative indices such as lesion-to-liver or lesion-to-mediastinum ratios and established MIBG scoring systems are applied where relevant. Optional comparator scans, when performed, follow the same quantitative framework; for 18F-FDG, lean-body-mass-normalized SUVs and metabolic tumor volume/total lesion glycolysis are recommended, and for CXCR4, lesion-to-liver or lesion-to-blood pool ratios may be recorded to assist harmonization. Image interpretation is performed by two blinded readers with adjudication of discrepancies, and lesion mapping records locations by compartment, including primary tumor, nodal stations, bone and bone marrow, soft tissue, liver, lung, adrenal, and other sites.

The reference standard integrates histopathology, correlative cross-sectional imaging, and clinical follow-up to adjudicate lesion truth status. In cases of modality discordance, targeted biopsy or directed follow-up is prioritized when clinically appropriate to refine the composite reference standard.

Data are captured in a validated electronic data capture environment with role-based access controls and full audit trails. The database implements automated range checks, temporal consistency checks for dose and acquisition timestamps, cross-form logic for tracer-modality pairing and pediatric weight-based dosing, and site-level reconciliation of imaging metadata (for example, DICOM headers) with case report forms. When optional comparator scans are performed, additional fields capture FDG-specific variables (fasting duration, pre-injection blood glucose, insulin use and timing, uptake time, ambient warming status) and CXCR4-specific variables (recent growth factor exposure and timing, white blood cell/absolute neutrophil counts when available, and timing of cytotoxic or steroid therapy relative to imaging). Source data verification is conducted on a predefined fraction of cases against medical records, radiopharmacy logs, imaging archives, and pathology reports. A comprehensive data dictionary specifies variable definitions, sources, units, coding standards such as MedDRA for adverse events, and normal or reference ranges where applicable. Written standard operating procedures govern study operations, including screening and consent, patient preparation and tracer administration, acquisition and reconstruction parameters, image reading and adjudication, data entry and query resolution, adverse event reporting, change control, and archival.

The study is exploratory in size and designed to estimate diagnostic performance with acceptable precision rather than to test a formal hypothesis. Primary analyses focus on SSTR- and NET-based imaging and will report per-patient and per-lesion sensitivity, specificity, accuracy, positive predictive value, and negative predictive value against the reference standard. Secondary and exploratory objectives include comparative effectiveness between NET and SSTR classes and within-class comparisons where intra- or inter-patient data allow, as well as subgroup analyses by disease category, metastatic distribution, and prior therapy. Where optional comparator scans are available, incremental and added-value analyses will evaluate their yield beyond SSTR/NET imaging using paired methods (for example, McNemar tests for sensitivity/specificity and decision-impact rates where management recommendations are captured). Statistical methods include exact confidence intervals for proportions, receiver operating characteristic analysis with area under the curve estimation, agreement metrics such as Cohen's kappa, and models that account for lesion-level clustering, for example generalized estimating equations. Multiplicity will be managed via hierarchical analysis plans or false discovery rate control for exploratory endpoints. Missing data are minimized prospectively through time-stamped workflows and automated completeness checks; missingness is categorized as missing, unavailable, non-reported, or not interpretable, and the primary analyses use complete-case datasets with sensitivity analyses employing appropriate imputation strategies when assumptions are defensible.

Safety oversight includes systematic collection of adverse events from tracer administration through follow-up, graded according to CTCAE version 5.0, with expedited reporting for serious and unexpected events per institutional and regulatory requirements. Radiation dosimetry is tracked at the participant level by tracer and modality, and cumulative exposure is maintained within diagnostic reference levels for the relevant age group. For optional comparator imaging, risks specific to the agents used are monitored and managed per protocol and local policy. The study is conducted in accordance with ICH-GCP and the Declaration of Helsinki, with institutional review board approval and written informed consent or assent obtained prior to any study procedures. Periodic monitoring and audits, on-site or remote as appropriate, verify adherence to the protocol, standard operating procedures, and the predefined data quality plan.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥6 months (pediatric and adult).
* Suspected or confirmed diagnosis of neuroblastoma (NB) or pheochromocytoma/paraganglioma (PPGL).
* Clinical indication for SSTR and/or NET-targeted molecular imaging for initial staging, restaging, suspected recurrence, response assessment, or treatment planning.
* Ability to undergo PET/CT or PET/MRI and/or SPECT/CT per protocol; for the PET/MRI subset, no MRI contraindications.
* Provision of written informed consent/assent per local regulations.
* Women of childbearing potential: negative pregnancy test within 72 hours prior to tracer administration and agreement to use effective contraception during the imaging window.
* For the multi-tracer subset (if applicable): willingness to undergo two imaging studies within a predefined window (e.g., ≤28 days) without intervening antitumor therapy.

Exclusion Criteria:

* Pregnant or breastfeeding; breastfeeding participants unwilling to follow tracer-specific lactation interruption guidance per institutional policy.
* Any condition that, in the investigator's judgment, precludes safe imaging or protocol compliance (e.g., uncontrolled cardiorespiratory disease, severe claustrophobia not amenable to sedation/anxiolysis).
* Known hypersensitivity to study radiopharmaceuticals or their excipients.
* Use of interfering medications without feasible washout:

NET imaging: drugs that affect catecholamine transport/storage (e.g., labetalol, tricyclic antidepressants, certain sympathomimetics) per site SOPs.

SSTR imaging: long-acting somatostatin analogues within ~3-4 weeks or short-acting within ~24-48 hours, unless clinically unavoidable.

* Prior therapeutic or high-dose 131I-MIBG within a period that would confound diagnostic imaging or dosimetry (e.g., within 6 months), at the investigator's discretion.
* Contraindications to required modality-specific procedures (e.g., MRI-incompatible implants for PET/MRI; iodinated/gadolinium contrast contraindication only if contrast is mandated and no alternative pathway is acceptable).
* Inability to lie still for the required acquisition time and sedation not feasible per institutional policy.
* Concurrent participation in an interventional study or receipt of anticancer therapy that would confound imaging interpretation within the imaging window; for multi-tracer comparisons, any interval systemic therapy between scans.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This single-center cohort comprises pediatric and adult patients with suspected or confirmed neuroblastoma (NB) or pheochromocytoma/paraganglioma (PPGL) who are referred for somatostatin receptor (SSTR) and/or norepinephrine transporter (NET)-targeted molecular imaging as part of diagnostic evaluation, staging, restaging, suspected recurrence assessment, response evaluation, or treatment planning (e.g., selection for peptide receptor radionuclide therapy or 131I-MIBG therapy). Participants are enrolled primarily from oncology, endocrinology, and nuclear medicine clinics of a tertiary academic medical center, with referrals from affiliated hospitals; most imaging is performed in the outpatient setting, with inpatient cases included when clinically indicated. Both sexes and all racial/ethnic groups are eligible, reflecting the catchment population.
  The study population includes a prespecified subset undergoing multi-tracer imaging when clinically justified and feasible, and a PET/MRI su
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
SUVmax | through study completion, an average of 1 year
  SUVmax is obtained by outlining a 3-D volume of interest (VOI) around the lesion on attenuation-corrected PET images; the software reports the single voxel with the highest activity concentration, normalized to injected tracer dose divided by the patient's body weight (MBq/kg).
SUVmean | through study completion, an average of 1 year
  SUVmean is obtained by outlining a 3-D volume-of-interest around the lesion on attenuation-corrected PET images and averaging all voxel values. Standardized uptake values are calculated as voxel activity concentration (kBq/mL) divided by injected activity per body weight (kBq/g).
Diagnostic Accuracy of SSTR and NET-Targeted Imaging | through study completion, an average of 1 year
  Per-patient and per-lesion sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and overall diagnostic accuracy compared to composite reference standard (histopathology when available and/or multidisciplinary clinical adjudication) Area under the receiver operating characteristic curve (AUC-ROC) for quantitative uptake metrics (SUVmax, SUVmean, target-to-background ratios)
Comparative Diagnostic Performance Between Tracer Classes | through study completion, an average of 1 year
  Head-to-head comparison of NET-targeted tracers (18F-MFBG, 123I-MIBG, others) versus SSTR-targeted tracers (68Ga-DOTA-peptides, 64Cu-DOTATATE, 18F-SSTR agents, others) in patients undergoing multi-tracer imaging Within-class comparative performance (e.g., 68Ga-DOTATATE vs 68Ga-DOTATOC vs 68Ga-DOTANOC; 18F-MFBG vs 123I-MIBG)

SECONDARY OUTCOMES:
Inter-reader Agreement | through study completion, an average of 1 year
  Cohen's kappa coefficient and percent agreement between two blinded readers for lesion detection and characterization Intraclass correlation coefficient for quantitative uptake measurements

CONTACTS AND LOCATIONS:
Overall Officials: Guoqiang Shao, Dr, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Within 6 months of the end of the trial, trial data are uploaded to http://www.medresman.org.cn/login.aspx
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 6 months and ending 3 years after the publication of results
Access Criteria: Qualified academic investigators with an IRB-approved proposal may request access to de-identified individual participant data (IPD), the full study protocol, blank case report forms, and the English/Chinese informed-consent templates. Requests should be emailed to the corresponding author; after signing a data-sharing agreement, files will be shared through a secure, password-protected institutional repository within 30 days.
URL: http://www.medresman.org.cn/login.aspx

REFERENCES:
- [Background] Gulaldi NCM, Gulleroglu NB, Cakmakci S, Gortan FA, Sari N. Dilemma on Pancreatic Uncinate Process Uptake on Ga68-DOTA Peptide PET/CT in Pediatric Neuroblastoma: Physiologic or Metastases? Curr Radiopharm. 2025;18(4):333-339. doi: 10.2174/0118744710226018250206105536. PMID 39966364
- [Background] Liu CJ, Ko KY, Lu MY, Hung WT, Chou SW, Du CJ, Chang HH, Hsu WM, Yang YL, Chien YT, Peng SS, Cheng MF. [68Ga]Ga-DOTA-TOC positron emission tomography outperforms [18F]FDOPA and [18F]FDG PET in pediatric neuroblastoma imaging: a prospective study. Eur J Nucl Med Mol Imaging. 2025 Dec;53(1):192-202. doi: 10.1007/s00259-025-07399-5. Epub 2025 Jun 13. PMID 40512254
- [Background] Lu Z, Sun Y, Zuo D, Li P, Sun X. Radiation Exposure to Patients and Others During Therapy for Pediatric Neuroblastoma With Lu-177-DOTATATE. Clin Nucl Med. 2025 Jun 1;50(6):480-485. doi: 10.1097/RLU.0000000000005763. Epub 2025 Feb 25. PMID 39992800
- [Background] Sharp SE, Trout AT, Weiss BD, Gelfand MJ. MIBG in Neuroblastoma Diagnostic Imaging and Therapy. Radiographics. 2016 Jan-Feb;36(1):258-78. doi: 10.1148/rg.2016150099. PMID 26761540
- [Background] Vik TA, Pfluger T, Kadota R, Castel V, Tulchinsky M, Farto JC, Heiba S, Serafini A, Tumeh S, Khutoryansky N, Jacobson AF. (123)I-mIBG scintigraphy in patients with known or suspected neuroblastoma: Results from a prospective multicenter trial. Pediatr Blood Cancer. 2009 Jul;52(7):784-90. doi: 10.1002/pbc.21932. PMID 19185008
- [Background] Giammarile F, Chiti A, Lassmann M, Brans B, Flux G; EANM. EANM procedure guidelines for 131I-meta-iodobenzylguanidine (131I-mIBG) therapy. Eur J Nucl Med Mol Imaging. 2008 May;35(5):1039-47. doi: 10.1007/s00259-008-0715-3. PMID 18274745
- [Background] Shulkin BL, Shapiro B. Current concepts on the diagnostic use of MIBG in children. J Nucl Med. 1998 Apr;39(4):679-88. PMID 9544682
- [Background] Leung A, Shapiro B, Hattner R, Kim E, de Kraker J, Ghazzar N, Hartmann O, Hoefnagel CA, Jamadar DA, Kloos R, Lizotte P, Lumbroso J, Rufini V, Shulkin BL, Sisson JC, Thein A, Troncone L. Specificity of radioiodinated MIBG for neural crest tumors in childhood. J Nucl Med. 1997 Sep;38(9):1352-7. PMID 9293786
- [Background] Bombardieri E, Giammarile F, Aktolun C, Baum RP, Bischof Delaloye A, Maffioli L, Moncayo R, Mortelmans L, Pepe G, Reske SN, Castellani MR, Chiti A; European Association for Nuclear Medicine. 131I/123I-metaiodobenzylguanidine (mIBG) scintigraphy: procedure guidelines for tumour imaging. Eur J Nucl Med Mol Imaging. 2010 Dec;37(12):2436-46. doi: 10.1007/s00259-010-1545-7. PMID 20644928
- [Background] Sharp SE, Shulkin BL, Gelfand MJ, Salisbury S, Furman WL. 123I-MIBG scintigraphy and 18F-FDG PET in neuroblastoma. J Nucl Med. 2009 Aug;50(8):1237-43. doi: 10.2967/jnumed.108.060467. Epub 2009 Jul 17. PMID 19617326